CLINICAL TRIAL: NCT06661200
Title: Exploratory Study of the Diagnostic Potential of an Innovative Thoracic Vibration Analysis Technique for Detecting Pulmonary and/or Cardiac
Brief Title: Exploratory Study of the Diagnostic Potential of an Innovative Thoracic Vibration Analysis Technique
Acronym: AIRFORCE2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-A02696-39
Record Dates: First submitted 2024-10-17; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-07

CONDITIONS: Cardiac Disease, Pulmonary Disease
Keywords: ultrasound, surface motion camera, sismography
MeSH Terms: conditions — Heart Diseases; Lung Diseases

STUDY DESIGN:
Intervention Model Description: Device feasability - Exploratory and feasibility study, monocentric, open, comparative, cross-sectional, made up of three groups:
  * cardiopathies (150 subjects)
  * healthy subjects (30 subjects)
  * pulmonary diseases (90 subjects)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy subjects N = 70 no cardiac and no pulmonary disease (Experimental): Healthy subjects who should undergo SMC recording after echocardiography and resporatory exploration.
  Interventions: Device: SMC signal recording
- Cardiac disease group (Experimental): Patients in this group had heart disease (n = 150): (i) aortic stenosis (ii) aortic leakage (iii) mitral leakage (iv) dilated cardimyopathy (v) or restrictive cardiomyopathy.
  Interventions: Device: SMC signal recording
- Respiratory failure (Experimental)
  Interventions: Device: SMC signal recording

INTERVENTIONS:
Device: SMC signal recording — SMC recording involves collecting vibrations from the thorax using an antenna equipped with piezoelectric crystals. Subjects face the machine or stand with their backs to the machine, shirtless. Acquisitions last around ten seconds.

SUMMARY:
Heart and lung disease are two major causes of hospitalisation and mortality in France (4-8). Together, these two diseases affect several million people in France, either acutely or chronically. They represent a major public health problem in social and economic terms.

Diagnosis of these disorders is often delayed, with acute decompensation preceded by a period of frustrating, non-specific clinical signs (9-12), which delay their discovery. Screening for these conditions in their early stages or diagnosing them in their acute form is crucial, but remains difficult because it requires multiple investigations that are costly and time-consuming (biology, radiology, ECG, etc.). The difficulty of diagnosis, the progressive profile and the ever-increasing frequency of these conditions (environmental and socio-economic factors) have considerably altered the landscape of medical emergencies and contributed to their difficulty.

The availability of a non-invasive technique capable of diagnosing both cardiac and pulmonary disorders without the help of an expert, without direct contact with the patient and without requiring his or her active participation, would be a major advance.

Technological innovations in all fields have always helped to improve patient care.The recent emergence of telemedicine and POCT(US) connected objects (point of care testing, point of care ultrasound)(13,14) is a good illustration of this.

A new technique using ultrasound, developed by the Langevin Institute (Surface Camera Motion) and supported by the start-up Austral Diagnostics, makes it possible, without direct contact with the subject, to record the propagation of thoracic vibrations induced by the functioning of the heart pump and respiratory mechanics.Consequently, any anomaly in the functioning of these organs can cause a change in the thoracic vibration regime and its propagation.

This completely new technique for exploring thoracic vibrations provides a particularly rich signal that has not yet been explored. Under these conditions, the signatures associated with cardiac and/or pulmonary pathologies are not yet perfectly defined.Furthermore, the diagnostic potential of this new technique in the early or acute phases of cardiopulmonary pathologies remains to be assessed.

In this prospective study, we propose to explore the signatures produced by this signal in various cardiac and respiratory pathologies.

The aim is To identify the discriminating criteria of the SMC signal that enable cardiac and pulmonary pathologies to be detected compared with a group of healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac disease OR respiratory failure OR healthy volunteer
* Affiliate to the social security system
* French-speaking
* Patient having been informed of the study and having signed informed

Exclusion Criteria:

* consent.BMI < 17 or BMI > 35
* Patients unable to stand for more than 10 minutes
* Patients unable to remain in apnea for 15 - 20 seconds
* Breast prosthesis wearers
* Wearers of pacemakers and/or defibrillators
* Valve prosthesis wearers
* Patients with difficulty understanding simple instructions (inspiration, expiration, respiratory blockage)
* Patients with severe hearing problems.
* Pregnant or breastfeeding woman. A urine pregnancy test will be performed if necessary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2025-02-14 (Estimated); Study Completion 2026-02-14 (Estimated)

PRIMARY OUTCOMES:
Surface Motion Camera (SMC) signal | baseline
  Identify the discriminating criteria of the SMC signal allowing the detection of cardiac pathologies on the one hand and pulmonary pathologies on the other hand versus a group of healthy subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided